CLINICAL TRIAL: NCT05739045
Title: A Multicenter, Prospective, Phase Ⅱ Clinical Study of Nivolumab Combined With SOX in the Perioperative Treatment of Locally Advanced Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Nivolumab Combined With SOX Used in the Perioperative Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiangdong Cheng (Other)
Responsible Party: Sponsor-Investigator, Xiangdong Cheng, Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stimulate-01
Record Dates: First submitted 2022-11-02; First posted 2023-02-22 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Immune Suppression; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nivolumab combined with SOX (Experimental): Medication regimen: nivolumab + SOX (3 cycles) before surgery → radical surgery (D2) → nivolumab + SOX (3 cycles) after surgery → nivolumab monotherapy maintenance (11 cycles); Surgery is performed 2 - 6 weeks after the last dose of neoadjuvant therapy, and postoperative adjuvant therapy is initiated at least 4 weeks after surgery.
  Interventions: Drug: nivolumab combined with SOX

INTERVENTIONS:
Drug: nivolumab combined with SOX — nivolumab + SOX (3 cycles) before surgery → radical surgery (D2) → nivolumab + SOX (3 cycles) after surgery → nivolumab monotherapy maintenance (11 cycles);

SUMMARY:
To evaluate the pathological complete response rate (pCR) of nivolumab combined with SOX (oxaliplatin + S-1) for neoadjuvant therapy of resectable gastric and gastroesophageal junction adenocarcinoma;

DETAILED DESCRIPTION:
Primary Objective

* To evaluate the pathological complete response rate (pCR) of nivolumab combined with SOX (oxaliplatin + S-1) for neoadjuvant therapy of resectable gastric and gastroesophageal junction adenocarcinoma; Secondary Objectives
* To evaluate the major pathological response rate (mPR), R0 resection rate, lymph node status after neoadjuvant therapy (ypN stage), 3-yr-DFS, OS, and safety and tolerability of nivolumab combined with SOX in the periopera; Exploration for markers of benefit groups

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be enrolled in the study:

1. Patients voluntarily participate in the study and sign the informed consent form; 2. Age ≥ 18 years and ≤ 75 years; 3. Have pathologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma; 4. Patients with gastric or gastroesophageal junction adenocarcinoma at the clinical staging of cT3-4 or N+, M0 (staging according to AJCC version 8) who could be radically resected as determined by CT and laparoscopy; 5. Have not received anti-tumor therapy (such as surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.); 6. Planned surgical treatment after completion of neoadjuvant therapy; 7. Able to swallow tablets normally; 8. ECOG score 0-1; 9. Expected survival >=12 months; 10. Main organ functions normal, i.e., meeting the criteria below:

1. Blood routine examination criteria shall meet:

   (No blood transfusion or blood products within 14 days, no G-CSF or other hematopoietic stimulating factors are used for correction) Absolute neutrophil count ≥1.5×109/L; Platelet ≥80×109/L; Hemoglobin ≥ 80 g/L
2. Criteria for biochemical tests:

Total bilirubin <1.5×ULN; ALT and AST≤2.5×ULN;

Serum Cr ≤ 1.5 × ULN or endogenous creatinine clearance > 50 ml/min (males: Endogenous creatinine clearance rate = ((140-age) × body weight)/(72 × serum Cr); female: endogenous creatinine clearance rate = ((140-age) × body weight)/(72 × serum Cr) × 0.85; body weight unit: kg; serum Cr unit: mg/mL):

11. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose and be willing to use a highly effective method of contraception during the trial and for 120 days after the last dose. Male subjects with partners of childbearing potential should be surgically sterilized or agree to use highly effective methods of contraception during the trial and for 120 days after the last dose;

Exclusion Criteria:

Patients with any of the following are not to be enrolled in the study:

1. Patients with unresectable factors, including unresectable tumor causes or unresectable surgical contraindications or refusal of surgery;
2. Previous or concurrent other malignancy;
3. Suffering from any chronic or major illness considered intolerable to treatment (eg, severe cardiac disease, uncontrolled hypertension, some degree of hepatic or renal dysfunction, etc.)
4. Patients who have previous gastrointestinal perforation, abdominal abscess or recent (within 3 months) intestinal obstruction or imaging and clinical symptoms suggestive of intestinal obstruction;
5. Patients having clinically significant bleeding symptoms or definite bleeding tendency within 3 months before the first dose of study drug, such as gastrointestinal bleeding, hemorrhagic gastric ulcer or suffering from vasculitis; if stool occult blood is positive at baseline, reexamination may be performed; if stool occult blood remains positive after reexamination, gastroscopy is required (except for patients having gastroscopy within 3 months before enrollment to exclude such condition);
6. Patients in the active stage of infection requiring treatment (such as antibacterial drugs, antiviral drugs, antifungal drugs);
7. Active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA ≥ 500 IU/ml; hepatitis C reference: HCV antibody positive and HCV viral copy number > upper limit of normal);
8. Patients with congenital or acquired immunodeficiency (such as HIV infection);
9. Patients with any active autoimmune disease or history of autoimmune disease with potential relapse;
10. Planned or previous organ or allogeneic bone marrow transplant;
11. Patients with current interstitial pneumonia or interstitial lung disease, or previous history of interstitial pneumonia or interstitial lung disease requiring steroids, or subjects with active pneumonia or severe lung function impairment on screening CT; active pulmonary tuberculosis;
12. Ongoing or recent treatment with immunosuppressive drugs or systemic corticosteroids to achieve immunosuppression;
13. Patients who have received a live attenuated vaccine within 28 days prior to the first dose of study drug or who require administration of such vaccine during treatment or within 60 days after the last dose;
14. Patients with known hypersensitivity to any of the study drugs or any of their excipients;
15. Nursing mothers;
16. Any factors that, in the judgment of the investigator, could affect patient safety and force the termination of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate (pCR) | 3 months
  pCR

SECONDARY OUTCOMES:
3-year DFS | 3 years
  3-year DFS

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Xiangdong, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Medication regimen: nivolumab + SOX (3 cycles) before surgery → radical surgery (D2) → nivolumab + SOX (3 cycles) after surgery → nivolumab monotherapy maintenance (11 cycles); Surgery is performed 2 - 6 weeks after the last dose of neoadjuvant therapy, and postoperative adjuvant therapy is initiated at least 4 weeks after surgery.
Supporting Information: Study Protocol